CLINICAL TRIAL: NCT00451022
Title: Follow-Up Study of Subjects Previously Enrolled in Immunotherapy Studies Utilizing Gene Transfer or Other Immunotherapeutic Agents
Brief Title: Follow-Up Study of Subjects Previously Enrolled in Poxviral Vector Gene Transfer Studies
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040274; 04-C-0274; NCT01444963 (obsolete NCT alias)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-03-28

CONDITIONS: Prostate Cancer; Liver Cancer; Breast Cancer; Colon Cancer; Lung Cancer
Keywords: Gene Therapy; Long Term Survivor; Research Specimen; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Liver Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects previously participating in gene transfer or other immunotherapy studies at the NCI or extramural sites receiving therapeutic agents as part of a multi-site trial.

SUMMARY:
This study aims to provide long-term follow-up care of patients previously enrolled in a vaccine study that involved poxviral vectors. Vectors are sequences of genetic material that can be used to introduce specific genes into genetic makeup. The study does not involve the use of any drug or biologic agent. Participants will undergo an annual health history. Because certain viruses enter into cells and create proteins from the viral genes, the type of vaccine treatment used is referred to gene therapy. The genes expressed by poxviral vectors do not become part of the genetic material left behind. Because gene therapy is a somewhat new technology, a prolonged monitoring of patients' health status is necessary, according to new specific reporting requirements for harmful events in patients who undergo such gene therapy studies. The risk of any long-term negative effects from the gene therapy that patients had received is quite small. Still, it is important that there be updates at least annually. This annual monitoring of health status will extend for 15 years, according to guidelines from the Food and Drug Administration, or for as long as patients are willing to participate.

Patients who received poxviral vectors (vaccinia or fowlpox, or both) at the National Cancer Institute, through a trial affiliated with the Laboratory of Tumor Immunology and Biology, may be eligible for this study.

Participants will be involved in the following forms of data collection:

* Annual medical history and physical examinations for the first 5 years following the last vaccine.
* Annual telephone contact during the last 10 years.
* Health status check, including primary cancer status, secondary malignancies, neurologic disorders, autoimmune disorders, and hematologic disorders.
* Blood tests for the presence of HIV antibodies.
* Reporting of medical problems, including information on unexpected hospitalizations and medications.

If a participant has died, the study will document the cause of death and autopsy information if available.

DETAILED DESCRIPTION:
This protocol aims to provide long-term follow-up and continued use of research specimens of participants previously enrolled on gene transfer or other immunotherapy studies at the National Cancer Institute as well as follow-up of subjects at extramural sites receiving these agents as part of a multi-site trial. Subjects will undergo an annual health history for up to 15 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who received poxviral vectors (vaccinia and/or fowlpox) or other vaccines utilizing gene transfer or any other immunotherapeutic agent through GMB, UOB and LTIB affiliated trials at the National Cancer Institute, as well as subjects at extramural sites receiving these agents as part of a multi-site trial. Available stored specimens obtained from NCI participants in GMB, UOB, and LTIB affiliated protocols may be transferred to this protocol for storage and eventual future research use.
* Subjects must be >= 18 years of age.

EXCLUSION CRITERIA:

Participants unwilling to participate.

(Please note, participants may participate in this protocol and, at the same time, participate in an active treatment or continuing care study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who received poxviral vectors (vaccinia and/or fowlpox) or other vaccines utilizing gene transfer or any other immunotherapeutic agent through GMB, UOB and LTIB affiliated trials at the National Cancer Institute, as well as subjects at extramural sites receiving these agents as part of a multi-site trial. These studies include (but are not limited to) the following NCI protocol numbers : 00-C-0137, 00-C-0154, 02-C-0218, 03-C-0176, 04-C-0167, 04-C-0246, 05-C-0017, 05-C-0167, 05-C-0229, 07-C-0106, 07-C-0107, 07-C-0188, 08-C-0166, 09-C-0101,11-C-0225, 12-C-0056, 13-C-0146, 13-C-0153, 13-C-0095, 14-C-0142, 14-C-0112, 15-C-020511-C-0247, 11-C-0262, 13-C-0063, 14-C-0090, 15-C-0012, 15-C-0118, 15-C-0145, 15-C-0178, 15-C-0179, 16-C-0035, 16-C-0048, 16-C-0079, 17-C-0007, 17-C-0023, 17-C-0038, 17-C-0057, and 17-C-0061.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2004-09-13 (Actual)

PRIMARY OUTCOMES:
To provide a mechanism for adequate follow-up of subjects previously participating in gene transfer or other immunotherapy studies at the National Cancer Institute as required by the U.S. Food and Drug Administration. | on-going
  Annual history and physical examinations for the first 5 years of follow-up and an annual telephone contact during the next 10 years.
To facilitate the continuous usage of stored research specimens collected from subjects under completed and ongoing protocols. | on-going
  Continued analysis on stored specimen samples until the samples are completely used.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Marte, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-C-0274.html